CLINICAL TRIAL: NCT02757157
Title: Determining the Metabolic Load of Walking in Water Compared to Walking on Land in People With COPD, Who Are Normal Weight and Obese, Compared to Peak Exercise Metabolic Response: a Prospective, Randomised Cross-over Pilot Trial
Brief Title: Comparison of Walking in Water and on Land in People With Chronic Obstructive Pulmonary Disease (COPD)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Hydrotherapy pool has closed.
Sponsor: European Respiratory Society (Other)
Collaborators: Center for Integrated Rehabilitation and Organ Failure Horn (Other)
Responsible Party: Principal Investigator, Renae McNamara, Clinical Specialist Physiotherapist, European Respiratory Society
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ERS STRTF 2015 - 9368
Record Dates: First submitted 2016-04-07; First posted 2016-04-29 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Hydrotherapy; Walking
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- COPD (normal weight) (Experimental): People with COPD (BMI 21 kg/m2 to 29 kg/m2)
  Interventions: Behavioral: Water-based walking; Behavioral: Land-based walking
- COPD (obese) (Experimental): People with COPD (BMI >/= 30 kg/m2)
  Interventions: Behavioral: Water-based walking; Behavioral: Land-based walking

INTERVENTIONS:
Behavioral: Water-based walking — Participants will walk in the water for 15 minutes at an intensity rating of five on the modified Borg scale for dyspnoea or perceived exertion, whichever is the highest. Walking intensity will be measured every three minutes during each walking session. If the intensity level is reported as below five, participants will be encouraged to increase the intensity by increasing their walking speed.
  During walking in water, VO2 and VE will be measured breath-by-breath using the Oxycon mobile. Every three minutes during the walking, heart rate, oxygen saturation, dyspnoea and exertion will be measured.
Behavioral: Land-based walking — Participants will walk on land for 15 minutes at an intensity rating of five on the modified Borg scale for dyspnoea or perceived exertion, whichever is the highest. Walking intensity will be measured every three minutes during each walking session. If the intensity level is reported as below five, participants will be encouraged to increase the intensity by increasing their walking speed.
  During walking on land, VO2 and VE will be measured breath-by-breath using the Oxycon mobile. Every three minutes during the walking, heart rate, oxygen saturation, dyspnoea and exertion will be measured.

SUMMARY:
The purpose of this study is to evaluate the metabolic load during a single session of moderate intensity walking in water compared to walking on land (over-ground) in people with chronic obstructive pulmonary disease (COPD) who are normal weight and obese, compared with peak exercise metabolic response.

The hypothesis is that the metabolic load of walking at a moderate intensity in water will be greater than walking on land.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of COPD (FEV1/FVC <0.7) in a clinically stable state (no acute exacerbation of COPD within the previous 4 weeks)
* accepting of walking in water
* BMI >/= 21 kg/m2

Exclusion Criteria:

* long-term oxygen therapy
* contraindications to entering a hydrotherapy pool

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-10; Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Breath-by-breath oxygen consumption (VO2) | Day of assessment during study measurement period (15 minutes)

SECONDARY OUTCOMES:
Minute ventilation (VE) | Day of assessment during study measurement period (15 minutes)

OTHER OUTCOMES:
Dyspnoea, measured by the modified Borg 0-10 category ratio scale | Day of assessment during study measurement period (15 minutes)
Exertion, measured by the modified Borg 0-10 category ratio scale | Day of assessment during study measurement period (15 minutes)
Oxygen saturation | Day of assessment during study measurement period (15 minutes)
Heart rate | Day of assessment during study measurement period (15 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Martijn A Spruit, PhD, Study Director — Centre of integrated rehabilitation for chronic organ failure
Locations (1):
- Centre of intergrated rehabilitation for chronic organ failure, Horn, Netherlands

IPD SHARING:
Plan to Share IPD: No